CLINICAL TRIAL: NCT04626037
Title: CLC Parent-Child Emotional Preparation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Einhorn Collaborative (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAT0109
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Emotional Connection; Child Development; Primary Prevention; Disruptive Behavior
Keywords: Welch Emotional Connection Screen (WECS) Toolkit; Nurture Science Program's (NSP); Children's Learning Centers (CLC); Parent-Child Emotional Preparation for Preschool
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Intervention Model Description: Using a pre-test, post-test design, this study will be comprised of a single group in which all participants are offered two Drop-In Zoom group sessions during the school semester.
  Exposure will vary at participant discretion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants in Group Zoom Sessions (Experimental): During each session, the mother-child dyads will meet with Nurture Science program staff virtually. The entire procedure will be done on Zoom or in person depending on school opening. All mother-child pairs will then be asked to interact, with the child sitting on the mother's lap face-to-face. The rest of the session may continue with: (1) Reading Cuddle and Calm Book (2) Mutual Mother and Child Emotional Exchange Prompts (3) Mothers Support Circle to identify and engage members of the mother's family in helping the dyad with emotional connection (4) Mommy Baby Book (5) Bottle of Emotions (6) Plans for continuing the work in the family. Returning mothers will be asked how they have progressed using the Cuddle and Calm and mutual narrative over the week and what their experience with their child after the session has been.
  Interventions: Behavioral: WECS Relational Toolkit

INTERVENTIONS:
Behavioral: WECS Relational Toolkit — The Cuddle and Calm Book, The Mommy Baby Book, mother and child mutual narrative, the Bottle of Emotions, and the WECS for emotional connection, make up the WECS Relational Health toolkit.

SUMMARY:
The purpose of this study is to investigate the feasibility of the Nurture Science Program's (NSP) Drop-In group via telemedicine as standard care at Children's Learning Centers (CLC) to prepare preschoolers emotionally for the preschool experience utilizing the Welch Emotional Connection Screen (WECS) Relational Health Toolkit. The behavioral, neurobiological, and clinical insights gained from this project may lead to better treatment of emotional, behavioral and developmental disorders.

DETAILED DESCRIPTION:
The purpose of this study is to test the practicality of mothers and children utilizing the WECS Relational Health Toolkit. The Cuddle and Calm Book, Well Baby Book, mother and child mutual narrative activity card, Bottle of Feelings, Mother's Socioemotional Support Circle, and the WECS for emotional connection make up the preschool WECS Relational Health toolkit. The WECS Relational Health Toolkit provides family-based resources to help mothers and children emotionally connect. The WECS Relational Health Toolkit is designed to create emotional connection and establish mother-child autonomic co-regulation, which helps shape autonomic state and behavior of the mother and child and therefore determines early child development and mother well-being. The investigators will test whether this toolkit can be a positive part of a standard preschool education program. Practicality will be measured through virtual participant attendance, a participant survey, and staff notes. Effects of this program on the emotional connection of mother-child pair will be measured through the Welch Emotional Connection Screen (WECS). Effects on child behaviors will be measured through the WECS-Parent Report (WECS-PR), SDQ, and Survey of Wellbeing of Young Children Baby Pediatric Symptom Checklist (BPSC) or the Preschool Pediatric Symptom Checklist (PPSC) subscales (age-dependent). We will also measure symptoms of depression in the mothers using the Center for Epidemiological Studies-Depression (CES-D) before and after the introduction to the Toolkit. We will also assess differences in developmental progress using the Milestones subscale of the SWYC.

ELIGIBILITY:
Inclusion Criteria:

- Preschool aged children from 0-5 years old and their mothers in CLC programs.

Exclusion Criteria:

- Families that choose not to participate in any data collection procedures but would like to listen in on the session(s).

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible dyads who enroll | 6 weeks
  This will be used to determine study uptake.
Proportion of participants who return for a second session | 6-12 weeks after first session
  This will be used to determine retention rate.

SECONDARY OUTCOMES:
Change in WECS screen scale score | 90 minutes (post-intervention); 6-12 weeks after first session; 6 months after first session
  Emotional connection will be measured from pre- and post-intervention WECS screen scale scores will be compared using paired sample t-tests. Change in WECS scores will be correlated with attendance using Spearman's rank correlation coefficient. This is a clinical tool completed by study staff to assess the emotional connection of a mother-child dyad. The WECS focuses on specific domains: attraction, vocal communication, facial communication, sensitivity/responsivity and one general: a dyad's interventional need. The WECS is scored based on observed presence of these 4 domains. The lowest score being a 1 and the highest being a 3. The higher the score, the more emotionally connected the dyad is therefore indicating a better outcome.

OTHER OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | 6 weeks post-intervention; 6 months after first session
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening questionnaire about 3-16 year olds. It exists in several versions to meet the needs of researchers, clinicians and educationalists. All versions of the SDQ ask about 25 attributes, some positive and others negative. These 25 items are divided between 5 scales: (1) emotional symptoms (5 items); (2) conduct problems (5 items); (3) hyperactivity/inattention (5 items); (4) peer relationship problems (5 items); (5) prosocial behavior (5 items). Sections (1) to (4) are added together to generate a total difficulties score (based on 20 items), ranging from 0 (better outcome) to 40 (worse outcome).
Survey of Wellbeing of Young Children (SWYC) Preschool Pediatric Symptom Checklist (PPSC) | 6-10 weeks after intervention, and again 6 months after first session
  The SWYC is a screening instrument for children up to 5 years of age. The Preschool Pediatric Symptom Checklist (PPSC) is used for children 18 months or older. Higher scores indicate higher risk.
Survey of Wellbeing of Young Children (SWYC) Baby Pediatric Symptom Checklist (BPSC) | 6-10 weeks after intervention, and again 6 months after first session
  The SWYC is a screening instrument for children up to 5 years of age. The Baby Pediatric Symptom Checklist (BPSC) is used for children under 18 months. Higher scores indicate higher risk.
Survey of Wellbeing of Young Children (SWYC) Milestones | 6-10 weeks after intervention, and again 6 months after first session
  The SWYC is a screening instrument for children up to 5 years of age. The Developmental Milestones (DM) of the SWYC will be used. Lower scores indicate higher risk.
Center for Epidemiologic Studies Depression Scale (CES-D) | 6-10 weeks after intervention, and again 6 months after first session
  The CES-D is a 20 item self-report inventory designed to assess current but nonspecific distress rather than clinically diagnosed depression.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Welch, MD, DFAPA, Principal Investigator — Columbia University
Locations (1):
- Childcare Learning Centers of Fairfield County, Stamford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided